CLINICAL TRIAL: NCT00806312
Title: The Expression and Significance of miRNA Profile and Markers of Inflammation in Patients With Pulmonary Arterial Hypertension
Brief Title: The Expression and Significance of MiRNA
Status: Completed | Type: Observational
Sponsor: Megan Ballinger (Other)
Responsible Party: Sponsor-Investigator, Megan Ballinger, Research Assistant Professor, Ohio State University
Organization: Ohio State University (Other)
Other Study IDs: 2008H0070
Record Dates: First submitted 2008-12-09; First posted 2008-12-10 (Estimated); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: MiRNA; pulmonary arterial hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1 PAH: Patients who are ≥ 18 years of age, not pregnant, and undergoing right heart catheterization for PAH diagnosis as part of their clinical care will be approached for consent and participation in this study.
- 2. Control: Patients who present with symptoms of PAH and whose clinical right heart catheterization doesn't support this diagnosis will be enrolled as control subjects.

SUMMARY:
It is not always known what causes PAH or what the best treatment is. The doctors doing this study would like to understand more about why some people develop PAH and other do not. They also would like to learn more about which treatments might help PAH and which people might respond better to treatments.

Doctors think that testing certain substances found in blood cells might help answer these questions. These substances are normally released by our bodies to protect us from infection and to tell the difference between normal and foreign substances in our body. Finally, a new test will study very small molecules called microRNA that control how our genes are expressed. This study is being done to see if blood samples can be tested to determine who might develop PAH, how well drugs will work to treat PAH and to learn more about the development of PAH.

DETAILED DESCRIPTION:
You will be asked to donate blood when you have your right heart catheterization and also at the 3-4 month follow-up visit. The amount of blood collected during your heart catheterization is about 20cc (about 4 teaspoons). This blood is discarded as part of the clinical catheterization procedure, but we are asking that we use it for this research study. Then, at the follow-up right heart catheterization, you will be asked to donate 20 cc (which is about 4 teaspoons) of blood.

If the second right heart is not required for clinical purposes then you will be asked to give a blood sample during your 3-4 month follow up clinic visit.

If you require an additional right heart catheterization, within one year, we will ask that you donate additional samples at the subsequent RHC.

Other data collected as part of your clinical care, such as medical history, chest x-ray (picture of your lungs), echocardiogram (picture of your heart), ventilation perfusion scan (determines how much blood goes to your lungs), chest CT (thin pictures of my lungs as slices), pulmonary function tests (breathing tests), and lab blood tests, will be used as part of this research.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* Not pregnant
* Undergoing right heart catheterization for PAH diagnosis

Exclusion Criteria:

* Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We expect to enroll 200 patients, who have been referred to the Pulmonary Hypertension Clinic at the Ohio State University Medical Center, in this study. Patients who are ≥ 18 years of age, not pregnant, and undergoing right heart catheterization for PAH diagnosis as part of their clinical care will be approached for consent and participation in this study.
Sampling Method: Non-Probability Sample
Enrollment: 207 (Actual)
Dates: Start 2008-07; Primary Completion 2018-08-16 (Actual); Study Completion 2018-08-16 (Actual)

PRIMARY OUTCOMES:
evaluate if miRNa profile and markers of inflammation in patients with PAH. These profiles may enable us differentiate patients that have PAH. This may assist in predicting response to therapy and enable us to optimize their treatment. may also shed s | end of study

CONTACTS AND LOCATIONS:
Overall Officials: Namita Sood, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States